CLINICAL TRIAL: NCT04631848
Title: ULTRASCORE™ Focused Force PTA Balloon Angioplasty for CLI Patients With Below the Knee Vessel Disease- a Multi-center Experience in 80 Subsequent Patients
Brief Title: ULTRASCORE™ Focused Force PTA Balloon Angioplasty for CLI Patients With Below the Knee Vessel Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Michael Lichtenberg, MD (Other)
Responsible Party: Sponsor-Investigator, Michael Lichtenberg, MD, Chief medical officer Vascular Center, Klinikum Arnsberg
Organization: Klinikum Arnsberg (Other)
Other Study IDs: ASL202001
Record Dates: First submitted 2020-11-06; First posted 2020-11-17 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Peripheral Arterial Disease (PAD)
Keywords: Scoring balloon dilatation
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ULTRASCORE™ Focused Force PTA Balloon
  Interventions: Device: ULTRASCORE™ Focused Force PTA Balloon

INTERVENTIONS:
Device: ULTRASCORE™ Focused Force PTA Balloon — The device will be used for percutaneous transluminal angioplasty (PTA) to dilatate calcified stenoses in below the knee vessels

SUMMARY:
The purpose of this single-arm, exploratory study is to evaluate safety and performance of treatment of critical limb ischemia (CLI) with the ULTRASCORE™ Focused Force balloon.

Patients with CLI in below the knee vessels will receive a percutaneous transluminal angioplasty with the device and will be followed up for 12 months.

DETAILED DESCRIPTION:
This single-arm, prospective, multi-center CE marked study (IIT) is planned to include up to 80 subjects with CLI in below the knee vessels with de novo stenoses or non-stented re-stenotic in total greater or equal 70% stenosis or occlusion of lower limb lesion. During the index procedure at Day 1 patients will be treated with ULTRASCORE™ Focused Force balloon.

Follow-up investigations for evaluation of parameters for primary and secondary endpoints will be performed at 4 weeks, 6 months, and 12 months after the index procedure..

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥ 18 years of age.
2. Patients are male or, if female, are either not of childbearing potential or must have a negative pregnancy test done within 7 days prior-index procedure and effective contraception must be used during participation in the Clinical Investigation.
3. Patients who are mentally and linguistically able to understand the aim of the Clinical Investigation and to show sufficient compliance in following the Clinical Investigation Plan.
4. Patients must agree to return for all required post-index procedure follow-up visits.
5. Patients are able to verbally acknowledge an understanding of the associated risks, benefits, and treatment alternatives to therapeutic options of the Clinical Investigation. Patients, by providing their informed consent, agree to these risks and benefits as stated in the patient informed consent document.
6. Rutherford Class 4-5
7. ≥70% stenosis of lower limb lesion by angio visual assessment
8. Target vessel(s) reconstitute(s) at or above the ankle with inline flow to at least one patent pedal vessel (includes perforating peroneal branches to dorsalis pedis and plantar artery).
9. The target lesion must either be de-novo or re-stenotic (stenosis ≥ 70% or occlusion by visual estimate). If the target lesion is re-stenotic, the prior PTA must have been done > 30 days prior-index procedure.
10. Treatment of multiple target lesions is allowed, as long as the composite target lesion length is ≤ 30 cm
11. At least one target lesion that is ≥ 2cm in length

Exclusion Criteria:

1. Patients with a known hypersensitivity or contraindication to aspirin, heparin, clopidogrel, or other anticoagulant/anti-platelet therapies, Paclitaxel (or analogs) or sensitivity to contrast media that cannot be adequately premedicated.
2. Patients with any contraindications as mentioned in the Instructions for Use (IFU) of the Investigational Device.
3. Patients with a life expectancy, from the Investigator's opinion, of less than 2 years.
4. Patients that are currently participating in other clinical investigations involving any investigational drug or device that may potentially confound the results of the Clinical Investigation, or that would limit the patient's compliance with the follow-up requirements of the Clinical Investigation.
5. Patients with a history of Myocardial Infarction (MI), thrombolysis or angina within 30 days prior-index procedure.
6. Patients with a history of major disabling stroke within 3 months prior index procedure.
7. Patients with a presence or history of severe renal failure (Glomerular Filtration Rate (GFR) ≤ 25 ml/min).
8. Patients who have undergone prior vascular surgery of the index limb to treat atherosclerotic disease.
9. Patients with clinically significant aneurysmal disease of the iliac, femoral or popliteal artery and patients with a history of clinically significant abdominal aortic aneurysm.
10. Target vessel(s) reconstitute(s) below the ankle with no inline flow to at least one patent pedal vessel.
11. Subjects scheduled to undergo a planned major amputation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from clinics with vascular centers
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Number of patients with patency of target lesion | 12 months
  Patency is defined as freedom from occluded target lesions (flow) verified by duplex ultrasound without re-intervention
Number of patients with composite safety | 4 weeks
  Freedom from major adverse limb events (MALE) and / or perioperative death

SECONDARY OUTCOMES:
Number of patients with patency measured with PSVR | 1, 6 and 12 months
  freedom from >50% restenosis in the target lesion as indicated by a duplex ultrasound peak systolic velocity ratio (PSVR) <2.5
Number of patients with secondary patency | 6 and 12 months
  freedom from occluded target lesions (flow) verified by duplex ultrasound
Number of patients with MAE (major adverse events) and MALE (Major adverse limb events) | 1 , 6 and 12 months
  composite of freedom from device- and procedure-related mortality, freedom from major target limb amputation and clinically driven TLR
Number of patients with procedural success | Day 1 after the index procedure
  ≤30% diameter stenose (DS) as determined by visual assessment
Number of patients with Device Success | Day 1 post Ultrascore usage
  ≤30% diameter stenose (DS) with no remaining flow limiting dissection as determined by visual assessment
Ankle-Brachial Index (ABI) | 6 and 12 months
Number of patients with Clinical success | 6 and 12 months
  improvement of at least one Rutherford class compared to the pre-procedure Rutherford classification
Number of patients with freedom from Target Lesion Revascularisation (TLR) | 6 and 12 months
Number of patients with freedom from Target Vessel Revascularisation (TVR) | 6 and 12 months
Number of patients with freedom from minor amputation | 6 and 12 months
Comparison of pain rating scale scores to Baseline | 6 and 12 months
  pain rating scale from 0 (no pain) to 10 (worst pain)
Comparison of the scores on the Walking Impairment Questionnaire (WIQ) to Baseline | 6 and 12 months
  individual scores for questions in the WIQ assessing the difficulties ranging from none (4) to not possible (0), Higher scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lichtenberg, Dr. med., Principal Investigator — Klinikum Hochsauerland GmbH
Locations (1):
- Klinikum Hochsauerland, Karolinen-Hospital, Arnsberg, Germany

IPD SHARING:
Plan to Share IPD: No